CLINICAL TRIAL: NCT02814006
Title: What is the Best Sexual Intercourse Strategy for Couples Actively Trying to Conceive?
Brief Title: Sexual Timing in Couples Actively Trying to Conceive
Acronym: SEXTACTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FPCEUP/RH3
Record Dates: First submitted 2016-06-17; First posted 2016-06-27 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2020-03

CONDITIONS: Conception
Keywords: marital relationship

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- every other day (Experimental): participants will visualize educational video with timed intercourse as recommended by NICE and ASRM
  Interventions: Other: health educational video
- fertile window (Experimental): participants will visualize educational video with timed intercourse as recommended by well-know evidence of better conception rates when using this strategy
  Interventions: Other: health educational video
- CG (No Intervention): participants will respond to questionnaire with no knowledge of intervention

INTERVENTIONS:
Other: health educational video — visualization of health educational video
  Arms: every other day; fertile window

SUMMARY:
This study will asses the effectiveness of two strategies for timed intercourse in couples actively trying to conceive

ELIGIBILITY:
Note: age limits are for female age only

Inclusion Criteria:

* Childless couples trying to conceive
* Relationship length > one year

Exclusion Criteria:

* Couples that already had achieved a successful pregnancy
* Couples with children

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in sexual functioning over the course of one year | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later]
  Self-report measure (FSFI, Rosen et al., 2000; IIEF, Rosen et al., 1997)

SECONDARY OUTCOMES:
Change in Depression over the course of one year | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later]
  Self-report measure (HADS, & Snaith Zigmund, 1994)
Change in Anxiety over the course of one year | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later]
  Self-report measure (HADS, & Snaith Zigmund, 1994)
Number of participants that attain an infertility diagnosis | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later]
Number of participants that achieve conception | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later]
Change in social support over the course of one year | T0 - before the intervention; T1 - one month later; T2 - six months later; T3 - one year later]
  Self-report measure (2WSS, Shakespeare-finch & Obst, 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana V Martins, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- University of Porto, Faculty of Psychology and Educational and Education Sciences, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martins MV, Fernandes J, Pedro J, Barros A, Xavier P, Schmidt L, Costa ME. Effects of trying to conceive using an every-other-day strategy versus fertile window monitoring on stress: a 12-month randomized controlled trial. Hum Reprod. 2022 Nov 24;37(12):2845-2855. doi: 10.1093/humrep/deac228. PMID 36272105